CLINICAL TRIAL: NCT00477022
Title: The Effects of Vacuum-Compression Therapy on the Healing of Diabetic Foot Ulcers
Acronym: VCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 86-456
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Vacuum compression therapy; Stereology; Ulcer Area; Vasotrain; Random Controlled Trial.
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vasotrain-447

SUMMARY:
the objective of this study is to evaluate the impact of vacuum-compression effects of Vasotrain on the diabetic foot ulcers using stereological method based on Cavalieri's principle in diabetic patients.

DETAILED DESCRIPTION:
Diabetic foot ulcers are common and serious complications of chronic diabetes mellitus. The prevalence of foot ulcers among patients with diabetes is 15%. The length of hospital stay is approximately 60% longer among patients with foot ulcers, as compared with those without ulcers. Diabetic foot ulcers accounts for >50% of all nontraumatic lower-leg amputations.Although, current preventive methods and treatment modalities have been effective in healing foot ulcers, statistics show high incidence of foot ulcers and amputations in individuals with diabetes.On the other hand, only a few studies were performed on the effects of Vasotrain in healing diabetic foot ulcers. The use of the machine enhances the delivery of oxygen and nutrients to the area, which in turn, facilitate wound healing

ELIGIBILITY:
Inclusion Criteria:

* A diabetic foot ulcer corresponding to grade 2
* No history of deep venous thrombosis and no hemorrhage in ulcer

Exclusion Criteria:

* Significant loss of protective sensation
* Hemorrhage during treatment
* Vertigo
* No completion of treatment

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Foot ulcer surface area was estimated stereologically, based on Cavalieri's principle before and after intervention, at pre treatment and post treatment | Baseline, 3 Weeks,

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Akbari, PhD, Principal Investigator — Deputy of research, Zahedan university of medical scinces
Locations (1):
- Dept. of physiotherapy, Zahedan university of medical scinces, Zahedan, Sistan & Bladchestan, Iran

REFERENCES:
- [Background] McCulloch JM Jr, Kemper CC. Vacuum-compression therapy for the treatment of an ischemic ulcer. Phys Ther. 1993 Mar;73(3):165-9. doi: 10.1093/ptj/73.3.165. PMID 8438004
- [Derived] Akbari A, Moodi H, Ghiasi F, Sagheb HM, Rashidi H. Effects of vacuum-compression therapy on healing of diabetic foot ulcers: randomized controlled trial. J Rehabil Res Dev. 2007;44(5):631-6. doi: 10.1682/jrrd.2007.01.0002. PMID 17943674
- See also: Provides extensive news and information about diabetes including symptoms, nutrition, weight loss, prevention, research, and community resources — http://www.diabetes.org